CLINICAL TRIAL: NCT01821196
Title: Density of Neurons in the Stomach and Prognosis of Gastric Adenocarcinoma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: due to insufficient quality of biopsy samples
Sponsor: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 210313
Record Dates: First submitted 2013-03-26; First posted 2013-03-29 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Stomach Neoplasms
Keywords: Tumor Markers, Biological; PGP9.5 protein, human; adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms; Adenocarcinoma | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- biopsy (Experimental): Additional biopsies by means endoscopy, 5 from tumor tissue, 5 from adjacent normal mucosa per patient.
  Interventions: Procedure: biopsy

INTERVENTIONS:
Procedure: biopsy — biopsies will be evaluated with immunohistochemistry and gene expression studies

SUMMARY:
Preclinical studies at our institution, based on a genetic mouse model of stomach cancer, strongly suggest that innervation of the stomach wall is deeply involved in tumorigenesis of stomach cancer. The data indicate that denervation of the stomach either by vagotomy or by injection of botulinum toxin (Botox®)in the stomach wall inhibits the development of cancer as well as reduces already established tumor volume in the stomach in this mouse model. Gene expression data indicate that vagotomy suppresses protein gene product 9.5 (PGP9.5). The expression of PGP9.5 is highly specific for the density of neurons and the diffuse neuroendocrine system. The investigators will take biopsies from tumors and adjacent normal mucosa either by means of endoscopy and/or from operative specimens from participants treated or evaluated for stomach cancer at the Department of Gastrointestinal Surgery, St Olavs Hospital, Trondheim University Hospital. The biopsies will be evaluated with immunohistochemistry and gene expression studies for the presence and density of PGP9.5. These data will be correlated to stage evaluation (TNM) and survival.

ELIGIBILITY:
Inclusion Criteria:

* Fifteen patients evaluated- or treated for suspected or verified gastric adenocarcinoma at the Department of Gastrointestinal Surgery, St Olavs Hospital, Trondheim University Hospital
* informed consent

Exclusion Criteria:

* General contraindications for endoscopy with biopsies (i.e. bleeding disorders or use of anticoagulants).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Density of PGP9.5 in gastric adenocarcinoma related to TNM stage and survival of stomach cancer | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jon Erik Grønbech, MD PhD, Principal Investigator — St. Olavs Hospital